CLINICAL TRIAL: NCT02690272
Title: " Expérience Vécue, Représentations et Processus Psychiques Chez Les Sujets en Attente de Transplantation Rénale "
Brief Title: "Lived Experience, Representations and Psychic Processes in Patients Awaiting Kidney Transplantation"
Acronym: LER-Psy-PAKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-A00971-48
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Kidney Tranplant
Keywords: kidney transplant; psychic process

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychic processes (Experimental): Quantitative and qualitative approche of the psychic process for patients awaiting kidney transplant
  Interventions: Behavioral: Psychic processes

INTERVENTIONS:
Behavioral: Psychic processes — Quantitative and qualitative aprroche of the psychic process

SUMMARY:
The kidney transplant remains the privileged treatment of the terminal renal insufficiency. This care is complex for the patient both on a medical surgical plan and by the psychic reorganizations. Among the temporary contraindications of transplantation, us retrouvonsdes psychological reasons. The research work consists in highlighting the psychic mechanisms of the subjects awaiting kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* stade 4 or 5 renal insufficiency
* Registered on waiting list for a first kidney transplant

Exclusion Criteria:

* in ward
* Unsigned consent
* Already transplanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-02-29; Primary Completion 2017-08 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Measure of anxiety | 6 months
  STAI-Y questionnaire with 20 items used to measure anxiety degree
Measure of psychic representations around transplant | 6 months
  ETA test: this test consists of an interview then the psychic projection through the drawing of 3 trees imagined by the patient and talking about him.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle COURTILLIE, Principal Investigator — University Hospital, Angers

REFERENCES:
- [Derived] Courtillie E, Fromage B, Augusto JF, Saulnier P, Subra JF, Bonnaud-Antignac A. Waiting for a kidney transplant, a source of unavoidable but reversible anxiety: a prospective pilot study investigating a psychological intervention. J Nephrol. 2023 Apr;36(3):841-849. doi: 10.1007/s40620-022-01535-2. Epub 2023 Jan 21. PMID 36670295